CLINICAL TRIAL: NCT01685255
Title: A Randomized, Open-Label, Phase 2 Study of the IDO Inhibitor Epacadostat Versus Tamoxifen for Subjects With Biochemical-Recurrent-Only Epithelial Ovarian Cancer, Primary Peritoneal Carcinoma, or Fallopian Tube Cancer Following Complete Remission With First-Line Chemotherapy
Brief Title: A Phase 2 Study of the IDO Inhibitor Epacadostat Versus Tamoxifen for Subjects With Biochemical-recurrent-only EOC, PPC or FTC Following Complete Remission With First-line Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated by the sponsor for lack of evidence of superiority and slow study accrual.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 24360-210
Record Dates: First submitted 2012-09-04; First posted 2012-09-14 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Ovarian Cancer; Genitourinary (GU) Tumors
Keywords: FIGO Stage III or IV EOC; PPC FTC; increasing CA 125
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms | interventions — epacadostat; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epacadostat (Active Comparator): Subjects randomized to Arm A (epacadostat) will take epacadostat tablets at a dose of 600 mg BID, beginning on Day 1.
  Interventions: Drug: Epacadostat
- Tamoxifen (Active Comparator): Subjects randomized to Arm B (tamoxifen) will take tamoxifen tablets at a dose of 20 mg BID, beginning on Day 1.
  Interventions: Drug: tamoxifen

INTERVENTIONS:
Drug: Epacadostat
  Other Names: INCB024360
  Arms: Epacadostat
Drug: tamoxifen
  Arms: Tamoxifen

SUMMARY:
This is an open-label, randomized, phase 2 study of an IDO inhibitor, INCB024360 (epacadostat) versus tamoxifen in biochemical recurrent only ovarian cancer patients following complete remission with first-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have received first-line chemotherapy, which must have been a platinum-containing regimen.
* Subjects who received maintenance paclitaxel or, bevacizumab, or alternative maintenance therapy (e.g. vaccines) are eligible for enrollment provided they have discontinued therapy at least 4 weeks for prior taxane and, at least 8 weeks for bevacizumab, or received medical monitor approval for time lapse from alternative maintenance therapy prior to randomization and recovered from toxicities to less than Grade 2.
* Subject must be currently in remission by clinical and radiological criteria (Response Evaluation Criteria for Solid Tumors [RECIST 1.1]).

  a. If a PET scan or high-resolution CT scan is performed and demonstrates new disease </= 1 cm, these subjects would be eligible.
* Clinical remission is defined as: asymptomatic and a negative physical examination.
* Scans are required post completion of platinum-containing therapy to document disease remission.
* Prior to the first-line regimen, CA 125 must have been elevated at first diagnosis, must have normalized with the first-line therapy/regimen, and is currently elevated:

  a. CA 125 elevation is defined as 2 consecutive measurements that are both above the Upper Limit of Normal (ULN) at least 42 weeks apart, with the second measure showing further increases from the first measurement
  1. If CA 125 is ≥ 2 × ULN the confirmatory value only needs to be 1 week apart.
  2. CA 125 elevation is defined as a value that is at least 2 × ULN on 2 occasions at least 1 week apart (UK ONLY REQUIREMENT).
* CA 125 elevation must be at least 3 months from completion of first-line platinum-containing regimen.
* Documentation of at least 1 normal CA 125 level at approximately 3 months during or following first line therapy is required.
* Subjects must have available archived tumor tissue.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate renal, hepatic, and bone marrow function based on screening laboratory assessments.

Exclusion Criteria:

* Subjects with any evidence of new disease (> 1 cm) including new ascites as confirmed by imaging.
* Any other prior antitumor systemic therapy except for first-line chemotherapy associated with previous CA 125 normalization or maintenance paclitaxel, bevacizumab, or alternative maintenance therapy as approved by the medical monitor.
* Subjects with prior radiotherapy within 3 months of randomization and have not recovered from all radiotherapy-related toxicities, who have received radiation therapy to the chest within 3 months of randomization, or who have a history or radiation pneumonitis.
* Subjects with protocol-specified active autoimmune processes except vitiligo or thyroiditis.
* Subjects receiving investigational study drug for any indication, immunological-based treatment for any reason (except completed adjuvant therapy with medical monitor approval), or potent CYP3A4 inducers or inhibitors.
* Subjects receiving monoamine oxidase inhibitors (MAOIs) within the 21 days prior to screening; subjects who have ever had Serotonin Syndrome (SS) after receiving 1 or more serotonergic drugs.
* Subjects for whom tamoxifen therapy is contraindicated.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2012-08; Primary Completion 2014-10-23 (Actual); Study Completion 2014-10-23 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) using Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 definition of progression as determined by the investigator. | PFS is defined as the number of days from randomization to the earlier of death or disease progression for up to 36 months.

SECONDARY OUTCOMES:
Safety and tolerability of epacadostat by adverse event assessment. | Adverse events assessed every 2 weeks during cycle 1, then every 28 days thereafter until each subject's death or disease progression or for up to 36 months, whichever is longest.
Cancer Antigen (CA) 125 response rate, using Gynaecologic Cancer Intergroup (GCIG) criteria. | CA 125 response rate defined as at least 50% reduction on study as compared to pretreatment sample; pre-treatment sample must be at least 2x ULN and response must be sustained for at least 28 days.
Duration of overall survival. | Overall survival followed every 12 weeks until last date known to be alive, until subjects withdraw consent or up to 36 months, whichever is longest.
Progression-free survival using RECIST 1.1 definition of objective progression as determined by the central imaging laboratory. | Progression free survival defined by central imaging lab using RECIST 1.1 assessed at 8 week intervals, retrospectively, until disease progression, death, subject withdraw of consent or up to 36 months, whichever is longest.

CONTACTS AND LOCATIONS:
Overall Officials: Lance Leopold, M.D., Study Director — Incyte Corporation
Locations (49):
- United States (17):
  - La Jolla, California
  - Los Angeles, California
  - San Francisco, California
  - Evanston, Illinois
  - Joliet, Illinois
  - Iowa City, Iowa
  - Covington, Louisiana
  - Baltimore, Maryland
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Bridgewater, New York
  - Buffalo, New York
  - Mineola, New York
  - Durham, North Carolina
  - Abington, Pennsylvania
  - Philadelphia, Pennsylvania
  - Greenville, South Carolina
- Australia (5):
  - Bendigo
  - Heidelberg
  - Herston
  - Milton
  - Randwick
- Canada (3):
  - Calgary, Alberta
  - Toronto, Ontario
  - Montreal, Quebec
- Russia (8):
  - Izhevsk
  - Krasnodar
  - Kursk
  - Moscow
  - Orenburg
  - Saint Petersburg
  - Ufa
  - Yekaterinburg
- Ukraine (4):
  - Chernivtsi
  - Dnipro
  - Kharkiv
  - Lutsk
- United Kingdom (12):
  - Bebington
  - Cardiff
  - Edinburgh
  - Glasgow
  - Keighley
  - Leeds
  - Liverpool
  - London
  - Manchester
  - Nottingham
  - Oxford
  - West Midlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kristeleit R, Davidenko I, Shirinkin V, El-Khouly F, Bondarenko I, Goodheart MJ, Gorbunova V, Penning CA, Shi JG, Liu X, Newton RC, Zhao Y, Maleski J, Leopold L, Schilder RJ. A randomised, open-label, phase 2 study of the IDO1 inhibitor epacadostat (INCB024360) versus tamoxifen as therapy for biochemically recurrent (CA-125 relapse)-only epithelial ovarian cancer, primary peritoneal carcinoma, or fallopian tube cancer. Gynecol Oncol. 2017 Sep;146(3):484-490. doi: 10.1016/j.ygyno.2017.07.005. Epub 2017 Jul 8. PMID 28698009